CLINICAL TRIAL: NCT06197932
Title: Effects of Big Toe Strength Training on Athletic Performance Parameter in Runners
Brief Title: Big Toe Strength Training on Athletic Performance Parameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/09
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Resistance Training; Athletic Performance; Running
Keywords: Big toe strengthening; Runners; Athletic performance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor) the assessor who will take the readings is blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine exercise and running training (Other): 15 participants were in experimental group giving them Toe strengthening exercise protocol along with running training for three weeks, measure all values before giving them protocol and after protocol. In pre measurements I assessed the strength of big toe of right and left feet, using the hip and toe dynamometer in kilograms. Further I assessed height of vertical jump in centimeters, than I assessed horizontal jump in centimeters. For balance Y -balance test is measured, test is measured for agility T test I measured, after assessment of all variables I gave them plan for big toe strengthening ask them to do repetitions about 15 in three sets twice a day, for 4 weeks after pre measurements, with intensity should be moderate. Asked them to perform 5 exercises twice a day. After 4 weeks measured all variable in same units and used the same instruments that used in pre measurements.
  Interventions: Other: Routine exercise and running training
- Big Toe Strengthening Exercise (Experimental): Pre-assessment measurements included big toe strength, vertical and horizontal jump heights, Y-balance for balance, and T-tests for agility. Following pre-assessment, participants followed a structured toe-strengthening protocol, performing 15 repetitions in three sets twice a day for 4 weeks. Post-intervention measurements, using the same units and instruments, aim to reveal the effects of the intervention on specified physical variables. This research provides insights into the potential benefits of combining toe-strengthening exercises with running training for enhanced physical performance.
  Interventions: Other: Big Toe Strengthening Exercise

INTERVENTIONS:
Other: Routine exercise and running training — impact of a 4-week running training program on physical performance variables in a control group comprising 15 participants. The control group exclusively underwent running training, and measurements were taken for variables such as the strength of the big toe of both right and left feet using a hip and toe dynamometer (measured in kilograms). Additionally, assessments included vertical jump height and horizontal jump distance (both measured in centimeters), balance using the Y-balance test, and agility via the T-test. All measurements were conducted with standardized equipment, both before and after the training period. se physical performance indicators.
  Arms: Routine exercise and running training
Other: Big Toe Strengthening Exercise — impact of a 4-week intervention involving toe-strengthening exercises and concurrent running training on 15 participants. Pre-assessment measurements included big toe strength, vertical and horizontal jump heights, Y-balance for balance, and T-tests for agility. Following pre-assessment, participants followed a structured toe-strengthening protocol, performing 15 repetitions in three sets twice a day for three weeks. Post-intervention measurements, using the same units and instruments, aim to reveal the effects of the intervention on specified physical variables. This research provides insights into the potential benefits of combining toe-strengthening exercises with running training for enhanced physical performance.
  Arms: Big Toe Strengthening Exercise

SUMMARY:
Running form and technique have a direct influence on a runner's economy, and therefore small changes in specific running mechanics could be useful to improving running performance. The thumb plays an important role in the functionality of the foot. During standing, the big toe is more loaded than the head of the five metatarsals and the heel. In this study, it will aimed to examine the relationship of big toe strength with parameters that affect anaerobic athletic performance in runners. In this study, it will aim to examine the relationship of big toe strength with parameters that affect anaerobic athletic performance in runners such as vertical jump, horizontally jumping, strength, agility and speed.

The study design will be Randomized Controlled Trial. This study will be conducted in Pakistan Sports Board (PSB) Lahore. The study will be completed within the time duration of eight to ten months after the approval of synopsis. Sample size will be 30 subjects. Non-probability convenient sampling technique will be used to recruit the individuals for the study and then randomization will be done by lottery method to divide the individuals into 2 treatment groups. The experimental group is given big toe strengthening program for 4 weeks along with running training on other hand control group will do only their running training and after that measures their pre post values on SPSS 25.

DETAILED DESCRIPTION:
Overall performance, particularly in a very popular sports activity such as running, is typically influenced by the status of the musculoskeletal system and the level of training and conditioning of the biological structures. Any change in the musculoskeletal system's biomechanics, especially in the feet and ankles, will strongly influence the biomechanics of runners, possibly predisposing them to injuries. A thorough understanding of the effects of a therapeutic approach focused on feet biomechanics, on the strength and functionality of lower limb muscles will contribute to the adoption of more effective therapeutic and preventive strategies for runners. this study group consists of male runners between the ages of 18-28. The participants will consist of a total of 30 people, 15 of which were in the experimental group and 15 in the control group. Time of the Study: study was determined as 2 days a week for 4 weeks. During this period, exercise with resistance bands to improve the toe strength will apply to the experimental group together with running training. The control group continued their running training and general lower extremity strength during this time Content of the Study: Extension (up) and flexion (down) exercises for the big toe will apply to the experimental group on the thera-band. The exercise will be done in 3 sets and 10-15 repetitions. The athletes got on the platform and performed the exercise according to the instruction of the researcher. The researcher will determine the tempo of the repetition numbers. All participants will command at the same tempo, and the number of repetitions and rest between sets will adjust equally. Measurement of Height: The height measurements of the participants will make with the height measuring device/ inch tape in cm. Measurement of Body Weight: without shoes and clothes (shorts and t-shirts may be allowed) while keeping his/her balance. Weight will measure on a weight machine in kilograms (kg). Measurement of Big Toe Strength: The strength rate of the big toe will take by using the Baseline brand digital display hydraulic pinch meter manufactured in the USA. Athletes placed their feet on the ground prepared in accordance with the big toe and adjust their big toes according to the location of the pinch meter. During the measurement, athletes will ask to apply maximum force with their big toe. Strength measurements will be made on the athletes in the sitting position without any support. Dynamic balance measurements of the participants will take with the Y balance test. To examine the effect of this training on the athletic performance parameters (vertical jump, force, and dynamic balance) were determined. Primary Null Hypothesis: • There is no significant Role of training on the athletic performance parameters (vertical jump, force, and dynamic balance) Primary Alternative Hypothesis: ● There is significant Role of training on the athletic performance parameters (vertical jump, force, and dynamic balance) Beneficiary industry: Runner Athletes The performance measures are underdeveloped for runners in Pakistan. With the help of this instrument runners can measure the toe strength and can increase or decrease the quantity of specific training program. Impact on teaching / training / institutional capability / local industry etc: There is scientific evidence that training with measurements can improve the result and its efficacy so calculated force by toe dynamometer. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Runners
* Previous history Doing Running practice from 1year for 3-4 days in a week(40-60minutes per day)

Exclusion Criteria:

* Any neurological signs.
* Any lower limb trauma or history of fracture past 6 month
* Diabetic, Hypertension

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Jump | pre and 4 weeks post intervention
  measured by vertical jump
Balance | pre and 4 weeks post intervention
  measured by Y balance test
Strength | pre and 4 weeks post intervention
  measured by Toe/Hip Dynamometer
Agility | pre and 4 weeks post intervention
  measured by T test

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denadai BS, Greco CC. Could middle- and long-distance running performance of well-trained athletes be best predicted by the same aerobic parameters? Curr Res Physiol. 2022 Jun 23;5:265-269. doi: 10.1016/j.crphys.2022.06.006. eCollection 2022. PMID 35800136
- [Background] Kurihara T, Terada M, Numasawa S, Kusagawa Y, Maeo S, Kanehisa H, Isaka T. Effects of age and sex on association between toe muscular strength and vertical jump performance in adolescent populations. PLoS One. 2021 Dec 31;16(12):e0262100. doi: 10.1371/journal.pone.0262100. eCollection 2021. PMID 34972181
- [Background] Yamauchi J, Koyama K. The mechanical role of the metatarsophalangeal joint in human jumping. PLoS One. 2022 May 20;17(5):e0268634. doi: 10.1371/journal.pone.0268634. eCollection 2022. PMID 35594285
- [Background] Yamauchi J, Koyama K. Importance of toe flexor strength in vertical jump performance. J Biomech. 2020 May 7;104:109719. doi: 10.1016/j.jbiomech.2020.109719. Epub 2020 Feb 26. PMID 32173032
- [Background] Shin H, Moon SW, Kim GS, Park JD, Kim JH, Jung MJ, Yoon CH, Lee ES, Oh MK. Reliability of the pinch strength with digitalized pinch dynamometer. Ann Rehabil Med. 2012 Jun;36(3):394-9. doi: 10.5535/arm.2012.36.3.394. Epub 2012 Jun 30. PMID 22837976
- [Background] Dobbs CW, Gill ND, Smart DJ, McGuigan MR. Relationship between vertical and horizontal jump variables and muscular performance in athletes. J Strength Cond Res. 2015 Mar;29(3):661-71. doi: 10.1519/JSC.0000000000000694. PMID 25226312